CLINICAL TRIAL: NCT04540718
Title: The Effects of Using Sauna Exposure to Augment Regular Exercise on Vascular Health and Hemodynamics
Brief Title: Exercise and Sauna on Blood Pressure and Cardiovascular Health
Acronym: ES2019
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jyvaskyla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UJyvaskyla
Record Dates: First submitted 2019-12-16; First posted 2020-09-07 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Cardiovascular Risk Factor; Heat Stress; Sedentary Behavior
MeSH Terms: conditions — Heat Stress Disorders; Sedentary Behavior | interventions — Exercise; Steam Bath

STUDY DESIGN:
Intervention Model Description: 3 groups of which; 1 serves as a control group, 1 exercise group, and 1 exercise and sauna group
Who Masked: Outcomes Assessor
Masking Description: Data statisticians (2) are blind to participant allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Participants in this group continues with their sedentary behavior
- Exercise only (Active Comparator): Participants in this group performs exercise 3 times a week (150 minutes total) according to the recommended exercise guidelines and will sit in the exercise laboratory for 15 minutes whilst the experimental group uses the sauna.
  Interventions: Other: Exercise
- Exercise and sauna (Experimental): Participants in this group performs exercise 3 times a week (150 minutes total) according to the recommended exercise guidelines and incorporates sauna bathing (heat therapy) immediately after exercise.
  Interventions: Other: Exercise; Other: Sauna

INTERVENTIONS:
Other: Exercise — 50 minutes of exercise, consisting of 20 minutes of resistance followed by 30 minutes of aerobic, three times a week for eight weeks.
  Other Names: Exercise training
  Arms: Exercise and sauna; Exercise only
Other: Sauna — 15 minutes of sauna exposure immediately after exercise intervention, three times a week for eight weeks.
  Other Names: Sauna bathing; Sauna exposure
  Arms: Exercise and sauna

SUMMARY:
The study aims to investigate the effects of including regular heat therapy when included to exercise. Specifically, participants in the sauna intervention group will undergo 15 minutes of sauna exposure immediately after a 50-minute session of exercise, 3 times a week, while participants in the exercise intervention group will follow only the same exercise protocol.

The 50-minute exercise session consists of 20 minutes of moderate intensity strength exercise, followed by 30 minutes of moderate-vigorous aerobic exercise on stationary bikes. This exercise intervention protocol was selected in order to meet and adhere to the recommended physical activity guidelines.

DETAILED DESCRIPTION:
The main purpose of the experiment is to investigate the cardiovascular modulations of sauna use with respect to vascular compliance and hemodynamics. The investigators seek to understand the long-term adaptations of regular sauna bathing in conjunction with exercise, particularly in sedentary populations with cardiovascular risk factors.

Of particular interests are the cardiovascular adaptations of regular sauna bathing when used in conjunction with exercise training; which meets the recommended minimum of current physical activity guidelines. Recent studies have shown that long-term sauna use with exercise is more effective than sauna use alone in patients with chronic heart failure. However several questions pertaining to regular exercise in combination with sauna use remain to be answered, as experimental data in the general population is still lacking.

This research project aims to find out the differences (if any) in cardiovascular and hemodynamic-related outcome parameters, between regular exercise according to the minimum recommended guidelines, and the same exercise program with an additional regular 15 minute sauna session post exercise.

The training intervention will last for 8 weeks, with each session consisting of 20 minutes of moderate intensity resistance training, followed by 30 minutes of aerobic training. Participants in the exercise only group rested in the training area for 15 minutes while the exercise and sauna participants went to the sauna for 15 minutes.

Temperature of the sauna room was increased by 5 degrees celsius every fortnight starting from 65 degrees celsius; during the final 2 weeks of the intervention the sauna temperature was at 80 degrees celsius. (65, 70, 75, 80). Participants were told that they could leave the sauna room anytime they felt uncomfortable or if they wish to.

ELIGIBILITY:
Inclusion Criteria:

* At least one conventional cardiovascular risk factor but asymptomatic for coronary heart disease or diabetes

Exclusion Criteria:

* Use of sauna more than once a week,
* Exercise more than 30 minutes a week,
* low blood pressure,
* any diagnosed and/or symptomatic cardiovascular disease,
* musculoskeletal injury,
* any other physical or mental condition that will prohibit the participation in the experiment,
* participation to any other study at the same time.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Hemodynamics | 8 weeks
  Blood pressure (systolic and diastolic)
Cardiovascular fitness | 8 weeks
  Estimated oxygen uptake

SECONDARY OUTCOMES:
Blood biomarker | 8 weeks
  Blood cholesterol (fasted)
Cardiac marker | 8 weeks
  Augmentation Index
Arterial stiffness | 8 weeks
  Pulse wave velocity
Body fat | 8 weeks
  Fat mass in kilograms

OTHER OUTCOMES:
Heart rate variability (HRV) | 8 weeks
  Heart rate variability
Haemoglobin concentration (endothelial function) | 8 weeks
  Moor instrument (moorVMS) near infrared spectroscopy (NIRS) will be used with a post occlusive reactive hyperaemia (PORH) protocol to assess haemoglobin concentration.
  The moorVMS-NIRS uses the established spatially resolved spectroscopy technique to measure absolute concentrations of oxygenated haemoglobin in human tissue. The system measures oxygenation using a probe which is placed in contact with the skin. Each probe consists of a detector head which contains two identical photodiodes and an emitter head which contains two near infrared light emitting diodes (LED) emitting light at approximately 750nm and 850nm. Light from the emitter head enters the tissue where it is subject to scattering and absorption. A small proportion of the incident light passes through the tissue to the photodiodes. The resulting photocurrents are amplified and acquired by the instrument.
Blood flow (endothelial function) | 8 weeks
  Moor instrument (moorVMS) laser doppler flowmetry (LDF) will be used with a post occlusive reactive hyperaemia (PORH) protocol to assess bloodflow (flux).
  The moorVMS-LDF uses the laser doppler technique where a low power laser light is transmitted via an optic fibre to the tissue. The light is scattered by tissue and moving blood cells and its frequency is Doppler broadened. Some of the scattered light is collected by one or more optic fibres and transmitted to a photo detector. The resulting photo current is electronically processed to produce the laser Doppler flux (blood flow) signal. The average Doppler frequency shift is directly proportional to the average speed of the blood cells.
Concentration of Nicotinamide Adenine Dinucleotide (NAD) | 8 weeks
  Nicotinamide Adenine Dinucleotide as measured from blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Jari A Laukkanen, PhD, Principal Investigator — University of Jyvaskyla
Locations (1):
- University of Jyväskylä, Jyväskylä, Central Finland, Finland

IPD SHARING:
Plan to Share IPD: No